CLINICAL TRIAL: NCT00612365
Title: Abdominal Body Composition, Inflammation, and Cardiovascular Disease
Brief Title: Association Between Abdominal Body Composition, Inflammation, and Risk for Cardiovascular Disease (The MESA ABD Study)
Acronym: MESA ABD
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Matthew A. Allison, University of California San Diego
Other Study IDs: 1419; R01HL088451 (NIH)
Record Dates: First submitted 2008-02-07; First posted 2008-02-11 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-02

CONDITIONS: Cardiovascular Diseases; Obesity
Keywords: Body Composition; Abdomen; Atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Participants from the Multi-Ethnic Study of Atherosclerosis (MESA) for abdominal aortic calcium (AAC) who have undergone computed tomography (CT) scans of the abdomen

SUMMARY:
Obesity is a growing public health concern, with approximately 31% of Americans considered obese. The link between abdominal obesity and cardiovascular disease (CVD) has been well established, but the effect of distinct types of abdominal fat tissue on CVD risk is not well known. The rate of obesity and the distribution of abdominal fat differ with age, sex, and ethnicity. These differences may have important implications for determining ethnic-specific relationships between abdominal body composition (ABC), inflammation, and CVD events. This study will evaluate the association between measures of abdominal fat, CVD risk, and inflammation in terms of ethnicity-, sex-, and age-specific differences.

DETAILED DESCRIPTION:
Abdominal obesity is a serious condition and increases the risk for potentially life-threatening cardiovascular diseases (CVDs). Abdominal fat is made up of structurally and functionally different tissues, which include visceral fat, subcutaneous fat, and intramuscular fat. The distribution and levels of these fat tissues are highly variable among obese people, and the effects of ABC differences on cardiovascular health are not well known. Notably, the standard measure of body mass index cannot distinguish between different kinds or ratios of tissue types that make up body weight and, therefore, may not be the best measurement tool. Determining the specific measures of these tissue types by computed tomography (CT) may provide better insight into the varied CVD risk seen among different ethnicities, sexes, and ages. This study will evaluate the association between volumetric measures of ABC, CVD risk, and inflammation in terms of ethnicity-, sex-, and age-specific variables.

This substudy will use data and specimens, including blood samples and CT scans, from participants in the Multi-Ethnic Study of Atherosclerosis (MESA) for abdominal aortic calcium (AAC). Stored blood samples will be used to perform assays for several measures of inflammation and to generate new data on biomarkers and subclinical CVD measures. The existing CT scans will be used to calculate five discrete volumetric measures of ABC, which will include subcutaneous fat, visceral fat, intramuscular fat, the visceral fat to visceral cavity ratio, and the lean muscle to visceral fat ratio. There will be no study visits for this study.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Inclusion Criteria:

* Participant in the MESA study

Exclusion Criteria:

* History of cardiovascualar disease

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will use data and specimens from participants in the MESA study for AAC who have undergone CT scans of the abdomen.
Sampling Method: Non-Probability Sample
Enrollment: 1975 (Actual)
Dates: Start 2007-09; Primary Completion 2012-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Relationship between abdominal tissue types, levels of inflammatory markers and adipokines, and CVD events | Measured at completion of sample analysis

SECONDARY OUTCOMES:
How differences in age, sex, and ethnicity influence the association between ABC and CVD risk | Measured at completion of sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A. Allison, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States